CLINICAL TRIAL: NCT03033914
Title: Phase I/II of Nivolumab and A(B)VD in the Front-line Setting for High Risk Hodgkin Lymphoma
Brief Title: A(B)VD Followed by Nivolumab as Frontline Therapy for Higher Risk Patients With Classical Hodgkin Lymphoma (HL)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry); Barbara Ann Karmanos Cancer Institute (Other); British Columbia Cancer Agency (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-1536; CA209-447 (Other: BMS)
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hodgkin Lymphoma
Keywords: Nivolumab; adriamycin; bleomycin; vinblastine; dacarbazine; 16-1536
MeSH Terms: conditions — Hodgkin Disease | interventions — Doxorubicin; Bleomycin; Vinblastine; Dacarbazine; Nivolumab

STUDY DESIGN:
Intervention Model Description: Cohort A will include patients less than 60 years of age with advanced stage (Stage III or IV) classical Hodgkin lymphoma (HL) who are at higer risk for relapse due to baseline international prognostic score (IPS) of 3-7 or positive PET scan after 2 cycles of ABVD (adriamycin, bleomycin, vinblastine, dacarbazine) ("PET-2 positive").
Masking Description: Cohort B will include patients 60 years of age and older with HL (any stage). AVD (adriamycin,vinblastine, dacarbazine)
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- < 60 years of age with advanced stage (HL) untreated (Experimental): The study will employ a 3+3 design and include 3 treatment cohorts. In each cohort, patients will receive 6 cycles of A(B)VD and 8 doses of nivolumab. In dose level 1, patients will receive nivolumab in combination with AVD during cycle 6 only followed by 6 additional doses of nivolumab. In subsequent dose levels, nivolumab will be combined with increasing numbers of cycles of AVD. Based upon safety data from another study with Nivolumab, we will no longer need to evaluate dose level 2. If we determine that dose level 1 is safe, the next group of patients will enroll onto dose level 3. A PET scan will be performed after 2 cycles of ABVD and those with a PET-negative response (defined by Deauville 1, 2 or 3) will proceed with 4 additional cycles of ABVD or AVD (per treating physician preference).
  Interventions: Drug: doxorubicin; Drug: Bleomycin; Drug: vinblastine; Drug: dacarbazine; Drug: Nivolumab
- 60 years of age and older with HL (any stage) untreated (Experimental): The study will employ a 3+3 design and include 3 treatment cohorts. In each cohort, patients will receive 6 cycles of AVD and 12 doses of nivolumab. In this cohort, patients will receive nivolumab in combination with AVD during cycles 5 and 6 only, followed by 8 additional doses of nivolumab. In subsequent cohorts, nivolumab will be combined with increasing numbers of cycles of AVD. Based upon safety data from another study with Nivolumab, we will no longer need to evaluate dose level 2. If we determine that dose level 1 is safe, the next group of patients will enroll onto dose level 3. Prophylactic growth factor support is mandatory for all patients on Cohort B and should be used per the treating physician's discretion for all other patients.
  Interventions: Drug: doxorubicin; Drug: vinblastine; Drug: dacarbazine; Drug: Nivolumab

INTERVENTIONS:
Drug: doxorubicin — Doxorubicin: 25 mg/m^2 will be administered by IV infusion on Days 1 and 15 of each 28-day cycle
Drug: Bleomycin — Bleomycin: 10 units/m^2 will be administered by IV infusion on Days 1 and 15 of each 28-day cycle
  Arms: < 60 years of age with advanced stage (HL) untreated
Drug: vinblastine — Vinblastine: 6 mg/m^2 will be administered by IV infusion on Days 1 and 15 of each 28-day cycle
Drug: dacarbazine — Dacarbazine (DTIC): 375 mg/m^2 will be administered by IV infusion on Days 1 and 15 of each 28-day cycle.
Drug: Nivolumab — nivolumab 240mg q14 days

SUMMARY:
The aim of this study is to improve the chance of cure for people with higher risk Hodgkin lymphoma. The purpose of the Phase I study is to test any good and bad effects of the study drug called Nivolumab when combined with ABVD for the front-line treatment of HL.The purpose of this Phase II study is to test whether including nivolumab in treatment for untreated Hodgkin lymphoma can improve the chance of cure for patients with abnormal PET scans after 2 cycles of ABVD.

DETAILED DESCRIPTION:
The phase II portion of cohort A will enroll patients with untreated stage III or IV Hodgkin lymphoma. All patients will begin with 2 cycles of ABVD as standard of care treatment. A PET scan will be performed after 2 cycles of ABVD. Enrollment at MSK may occur at any point during the first two cycles of ABVD treatment. Enrollment at non-MSK locations will occur after the PET scan is performed. MSK patients with a PET-negative response (defined by Deauville 1, 2 or 3) will proceed with 4 additional cycles of ABVD or AVD (per treating physician preference) on-study. Non-MSK patients with a PET-negative response are not eligible for this study. Patients with a PET-positive response (Deauville 4 or 5) will proceed with 4 cycles of AVD plus nivolumab on-study. Non-MSK patients must have a PET-positive response to enroll on this study

ELIGIBILITY:
Inclusion Criteria:

* Cohort A overview: Patients age less than 60 with untreated stage III or IV classical Hodgkin lymphoma will be eligible for cohort A. In phase I, patients could enroll onto cohort A if they had have a baseline IPS ≥3 OR if their PET scan after 2 cycles of ABVD is positive (Deauville 4 or 5). Enrollment onto phase I has now ceased and enrollment will begin for phase II.

In phase II, patients less than 60 years of age with stage III or IV HL are eligible. MSK patients may enroll anytime within the first 2 cycles of ABVD Non-MSK patients must enroll after positive PET-2 scan.

* Cohort B overview: Patients 60 or older with untreated classical Hodgkin lymphoma (regardless of stage) will be eligible for cohort B.

The following eligibility criteria applies to both cohort A and B except when stated otherwise:

* Histologic diagnosis of classical Hodgkin lymphoma

  * FDG-avid disease by FDG-PET/CT
  * Non-MSK patients ONLY: PET-2 positive disease (Cohort A only)
  * Ann Arbor Stage III or IV disease (Cohort A only)
  * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 2 weeks prior to the start of study drug. Women who undergo fertility preservation within 2 weeks of beginning chemotherapy are expected to have false-positive pregnancy tests and therefore testing may be waived for these patients.
  * WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug. Women who undergo fertility preservation within 2 weeks of beginning chemotherapy are expected to have false-positive pregnancy tests and therefore testing may be waived for these patients.
  * Reliable methods of birth control include a double barrier method, oral contraceptive, implant, dermal contraception, long-term injectable contraceptive, intrauterine device, tubal ligation or total abstinence during the study
  * Women must not be breastfeeding
* Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (i.e. use of a condom during intercourse) for the duration of treatment with study drug plus 5 half-lives of study drug plus 90 days (duration of sperm turnover) for a total of 31 weeks posttreatment completion
* Age ≥ 18
* Serum creatinine ≤ 1.5 x Upper limit of normal (ULN) or creatinine clearance (CrCl) ≥ 40 mL/min (measured using the Cockcroft-Gault formula
* AST/ALT ≤ 3 x ULN (5x ULN for those with lymphoma involvement of the liver)
* Total bilirubin ≤ 1.5 x ULN (except subjects with Gilbert Syndrome, who can have total bilirubin < 3.0 mg/dL)

Exclusion Criteria:

* Subjects with active brain metastases or leptomeningeal metastases.
* Subjects with nodular lymphocyte-predominant HL
* Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
* Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
* Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Subjects with a condition requiring systemic treatment with systemic corticosteroids (equivalent of >10mg/day of prednisone). Patients may receive steroid therapy if steroids are tapered down to 10mg or less by 4 weeks after initiating A(B)VD to control lymphoma-related symptoms.
* Any of the following cardiovascular conditions or values within 6 months before the first dose of study drug:

  * A left-ventricular ejection fraction < 50%
  * Myocardial infarction within 2 years of randomization
  * New York Heart Association (NYHA) Class III or IV heart failure
* Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
* Any positive test for hepatitis B virus or hepatitis C virus indicating acute infection.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* History of severe hypersensitivity reaction to any monoclonal antibody.
* Adjusted DLCO <60% (if unadjusted DLCO is >/=60% then there is no need to calculate adjusted

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2017-01-25 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
number of patients who have dose limiting toxicity | 2 years
  For this objective, the standard 3+3 scheme will be used. Initially, 3 patients will enroll onto dose level 1. If no patients experience DLT, enrollment will proceed to the next dose level. If 1 DLT is observed, 3 additional patients will enroll onto dose level 1. If 1 or fewer patients out of 6 experience DLT, enrollment will proceed to the next dose level. If 2 or more DLTs are observed at a given dose level, the previous dose will be declared the MTD. Adverse events will be assessed according to the Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. If CTCAE grading does not exist for an adverse event, the severity of mild, moderate, severe, and life-threatening, corresponding to Grades 1 - 4, will be used.
Phase II- progression free survival | 2 year
  The updated response criteria entitled "The Lugano Classification" system will be applied to define complete response, partial response, and progression of disease in this study.

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (10):
- United States (9):
  - Karmanos Cancer Institute, Detroit, Michigan
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Hackensack Meridian Health, Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
- BC Cancer (Data Collection Only), Vancouver, Canada

REFERENCES:
- [Derived] Torka P, Feldman T, Savage KJ, Ganesan N, Drill E, Hancock H, Davey T, Perez L, Capadona C, Subzwari S, Galasso N, Yang J, Post M, Boardman A, Caron P, David K, Epstein-Peterson Z, Falchi L, Ghione P, Hamlin P, Horwitz SM, Intlekofer AM, Johnson W, Kumar A, Lue J, Noy A, Owens C, Palomba ML, Salles GA, Steiner R, Stuver R, Vardhana S, Yahalom J, Dogan A, Zelenetz AD, Schoder H, Moskowitz AJ. Phase II Trial of Nivolumab Plus Doxorubicin, Vinblastine, Dacarbazine as Frontline Therapy in Older Adults With Hodgkin Lymphoma. J Clin Oncol. 2025 Mar 10;43(8):985-993. doi: 10.1200/JCO-24-01278. Epub 2024 Dec 11. PMID 39661923
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm